CLINICAL TRIAL: NCT06590805
Title: Ameliorative Potential of Electroacupoint for Diminutive Milk Production in Lactating Woman
Brief Title: Electroacupoint for Diminutive Milk Production
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haytham Ibrahim Morsi (Other)
Responsible Party: Sponsor-Investigator, Haytham Ibrahim Morsi, Lecturer, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.1 993
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Physical Therapy; Electrotherapy; Dietary Modification
Keywords: Electroacupoint; Postnatal care; Diminutive milk production; Lactating woman
MeSH Terms: interventions — Iron

STUDY DESIGN:
Intervention Model Description: Two Parallel Groups for Comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electroacupoint combined with postnatal care (Experimental): Electroacupoint stimulation using the Electroacupoint device and postnatal care diet in form of balanced diet and drinking sufficient clean water and routine postnatal care.
  Interventions: Procedure: Electrotherapy using Chattanooga stimulation unit; Dietary Supplement: Balanced Diet using domperidone drug, iron, and folic acid supplementation.
- postnatal care only (Active Comparator): Postnatal care diet in form of balanced diet and drinking sufficient clean water and routine postnatal care.
  Interventions: Dietary Supplement: Balanced Diet using domperidone drug, iron, and folic acid supplementation.

INTERVENTIONS:
Procedure: Electrotherapy using Chattanooga stimulation unit — Electroacupoint stimulation using the Chattanooga intellect transport 2-channel electrotherapy stimulation unit 2783. It uses the influences energy flows by needling the acupuncture points which lie along the body meridians to achieve a harmonious balance between physical, emotional, and spiritual states. The same effect can be achieved without the use of needles. These needleless stimulations are noninvasive and nontraumatic and are useful for individuals who are scared of needles. They are also associated with decreased risk of infection or bruise.
  Arms: Electroacupoint combined with postnatal care
Dietary Supplement: Balanced Diet using domperidone drug, iron, and folic acid supplementation. — Postnatal care diet in form of balanced diet using domperidone drug, iron, and folic acid supplementation. Additionally, drinking sufficient clean water and routine postnatal care.
  It was performed by asking the participant to take ten mg domperidone three times a day after meals. Iron and folic acid supplementation were also continue for three months after birth.

SUMMARY:
The purpose of this study was to reveal the effect of electroacupoint on scanty milk production in lactating women.

DETAILED DESCRIPTION:
Postnatal scanty milk secretion is a common complaint. Some physical and medicinal therapies have been proposed to enhance milk production. These therapies must be both successful and safe for both the mother and the child. In many cases, milk supply can be increased by frequent, regular milk removal, Medication to increase milk supply (galactogogues) such as domperidone.

Domperidone has been linked to maternal adverse effects in galactogogue trials and cases reported to the Food and Drug Administration include dry mouth, headache, dizziness, nausea, abdominal cramping, diarrhea, palpitations malaise, and shortness of breath. Some of these were more frequent with dosages greater than with 30 mg daily. Drug withdrawal symptoms consisting of insomnia, anxiety, and tachycardia were reported in a woman taking 80 mg of domperidone daily for 8 months as a galactogogue who abruptly tapered the dose over 3 days.

ELIGIBILITY:
Inclusion Criteria:

* They were complaining of insufficiency of lactation within the first month after cesarean section.
* They are using mixed feeding; both breast and bottle feeding, between three and six bottles per day.
* Their age ranged from 25-30 years old.
* Their body mass index didn't exceeded 30 kg/m2.

Exclusion Criteria:

* Postpartum haemorrhage.
* Cardiorespiratory disease.
* Diabetes mellitus.
* Breast cancer.
* Previous surgeries in the chest, breast, or the surrounding area.
* Anemia.
* Any causes that hindered their normal breastfeeding (retraced, cracked, inflamed, or inverted nipples).
* Receiving contraceptive pills.
* Having infants with conditions that may affect the lactation process such as congenital abnormalities of the mouth (tongue tie, cleft palate).
* Congenital heart disease.

Ages: 25 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is specified for Females who have diminutive milk production.
Enrollment: 36 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Baby Weight. | Change from Baseline Baby Weight at three months.
  Measurement of Baby Weight using the Baby Weight Scale.
Change in Serum Prolactin Level. | Change from Baseline Serum Prolactin Level at three months.
  Measurement of Serum Prolactin Level using the Serum Blood Test.
Change in Flow of Milk. | Change from Baseline Flow of Milk at three months.
  Measurement of Flow of Milk using the Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Haytham I Morsi, M.Sc., Study Director — Kafrelsheikh University
Locations (1):
- Kafrelsheikh University, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No